CLINICAL TRIAL: NCT05160233
Title: Digital Treatments for Opioids and Other Substance Use Disorders (DIGITS) in Primary Care: A Hybrid Type-III Implementation Trial
Brief Title: Digital Treatments for Opioids and Other Substance Use Disorders in Primary Care
Acronym: DIGITS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1794767; R01DA047954 (NIH)
Record Dates: First submitted 2021-12-03; First posted 2021-12-16 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Drug Use Disorders; Illicit Drug Use; Alcohol-Related Disorders; Opioid Use Disorder
Keywords: substance use disorders; mHealth; digital therapeutics; primary care; implementation science; randomized controlled trial; factorial trial; opioid use disorders
MeSH Terms: conditions — Substance-Related Disorders; Alcohol-Related Disorders; Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Cluster-randomized trial with 2x2 factorial randomization of two experimental strategies resulting in four arms: 2x2 factorial design to four approaches: (1) "standard implementation"; (2) "standard implementation plus practice facilitation"; (3) "standard implementation plus health coach"; and (4) "standard implementation plus both.
Who Masked: Outcomes Assessor
Masking Description: All outcomes are derived from secondary administrative data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard Implementation (Active Comparator): All primary care clinics will implement reSET and reSET-O using standard implementation approach.
  Interventions: Behavioral: Standard implementation
- Standard Implementation Plus Health Coaching (Experimental): The clinics in this arm will implement reSET and reSET-O with a standard implementation strategy and patients at the clinic will receive support from a health coach to help them engage with reSET and reSET-O.
  Interventions: Behavioral: Standard implementation; Behavioral: Health Coaching
- Standard Implementation Plus Practice Facilitation (Experimental): The clinics in this arm will implement reSET and reSET-O with a standard implementation strategy and a practice facilitator will provide the clinic with support for implementation.
  Interventions: Behavioral: Standard implementation; Behavioral: Practice Facilitation
- Standard Implementation Plus Health Coaching and Practice Facilitation (Experimental): The clinics in this arm will implement reSET and reSET-O with a standard implementation strategy and patients at the clinic will receive support from a health coach to help them engage with reSET and reSET-O. Additionally, a practice facilitator will provide the clinic with support for implementation.
  Interventions: Behavioral: Standard implementation; Behavioral: Health Coaching; Behavioral: Practice Facilitation

INTERVENTIONS:
Behavioral: Standard implementation — Brief clinician training and an implementation toolkit consisting of job aids, patient educational materials, scripted conversations, electronic health record tools, and a population management workbench.
Behavioral: Health Coaching — The clinic is provided access to a health coach who conducts outreach with patients. The health coach facilitates engagement with the digital therapeutic and encourages contact with the care team.
  Arms: Standard Implementation Plus Health Coaching; Standard Implementation Plus Health Coaching and Practice Facilitation
Behavioral: Practice Facilitation — A trained facilitator provides support for implementation by delivering the following interventions to clinic staff: Bolster Education, Audit and Provide Feedback, Support Plan-Do-Study-Act Cycles, Engage Others in Change.
  Arms: Standard Implementation Plus Health Coaching and Practice Facilitation; Standard Implementation Plus Practice Facilitation

SUMMARY:
The DIGITS Trial addresses a critical knowledge gap: How to best implement digital treatments for opioids and other substance use disorders in primary care. The DIGITS Trial is a partnership between Kaiser Permanente Washington Health Research Institute (KPWHRI) in Seattle, and Kaiser Permanente Washington, a healthcare delivery system in Washington State.

In this study, the FDA-authorized reSET and reSET-O digital therapeutics will be implemented in Kaiser Permanente Washington primary care clinics. The study will evaluate the extent to which two implementation strategy interventions, health coaching and practice coaching, improve the implementation. Primary care clinics are randomized to receive these implementation strategy interventions. Each clinic will have a 12-month active implementation period beginning on its date of randomization. To study the continued use of reSET and reSET-O after the active implementation period is completed, a sustainment period of up 12 months will follow the active implementation period.

DETAILED DESCRIPTION:
Specific Aims of the DIGITS Trial are to:

1. Estimate the effect of practice facilitation and health coaching implementation strategies in increasing the reach and fidelity of a digital therapeutic for substance use disorders in primary care clinics.
2. Compare the population-level cost-effectiveness of each implementation strategy in increasing reach, fidelity, and abstinence.

ELIGIBILITY:
Patient Inclusion Criteria:

* Had a primary care visit in a participating clinic during the active implementation period or sustainment period
* Screened positive for substance use on the day of the visit or in the prior year
* Adult aged 18 years or older at time of visit

Clinic Inclusion Criteria:

- At least 1 clinician trained in the use of reSET/reSET-O

Patient Exclusion Criteria:

- Patients who have requested through their health system to opt out of research

Clinic Exclusion Criteria:

- Previously participated in a pilot implementation of reSET/reSET-O

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13000 (Estimated)
Dates: Start 2021-12-09 (Actual); Primary Completion 2024-09-09 (Estimated); Study Completion 2024-09-09 (Estimated)

PRIMARY OUTCOMES:
Reach of the digital therapeutic to patients in the primary care clinic | 12 months
  The proportion of patients who initiate the digital therapeutic, defined by instances in which patients open the app, enter the prescription code, and use a treatment module.
Fidelity of patients' use of the digital therapeutic to clinical recommendations | 15 months
  Mean number of weeks during patients' 12-week prescription in which patients use 4 app modules/week and have visited a clinician in the past 30 days

SECONDARY OUTCOMES:
Engagement | 15 months
  Mean number of months in which patients make ≥1 visit for substance use disorder
Economic costs | 12 months
  Costs from the perspective of a health system and payer including implementation, direct intervention, operating, and other indirect health care costs. This measure will be used to calculate the population-level cost effectiveness of increasing reach, fidelity, and engagement.

OTHER OUTCOMES:
Reach-2 | 12 months
  The proportion of patients prescribed reSET or reSET-O
Fidelity-2 | 15 months
  Mean number of weeks in which patients use at least 1 module/week
Sustainment | 12 months
  The proportion of patients who are reached during the sustainment period
Substance use | Up to 18 months from the patients index visit date
  The proportion of patients who are reached and reduce their substance use
Abstinence | Up to 18 months from the patients index visit date
  The proportion of patients who are reached and are abstinent from substances

CONTACTS AND LOCATIONS:
Overall Officials: Joseph E Glass, PhD, MSW, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wong ES, Dorsey CN, Beatty TC, Bobb JF, Stefanik-Guizlo K, Key DL, Ramaprasan A, Idu AE, Fortney JC, Mogk J, Palazzo L, Caldeiro RM, King D, McWethy AG, Glass JE. Economic cost of strategic implementation approaches to increase uptake of digital therapeutics for substance use disorders in a large integrated health system. PLOS Digit Health. 2026 Jan 8;5(1):e0001145. doi: 10.1371/journal.pdig.0001145. eCollection 2026 Jan. PMID 41505485
- [Derived] Glass JE, Dorsey CN, Beatty T, Bobb JF, Wong ES, Palazzo L, King D, Mogk J, Stefanik-Guizlo K, Idu A, Key D, Fortney JC, Thomas R, McWethy AG, Caldeiro RM, Bradley KA. Study protocol for a factorial-randomized controlled trial evaluating the implementation, costs, effectiveness, and sustainment of digital therapeutics for substance use disorder in primary care (DIGITS Trial). Implement Sci. 2023 Feb 1;18(1):3. doi: 10.1186/s13012-022-01258-9. PMID 36726127